CLINICAL TRIAL: NCT04460287
Title: Bioavailability of Different Formulas Enriched With DHA Using Wet Mixing or Dry Blending Method
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Indonesian Nutrition Association (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Basic Science
Other Study IDs: INA/NM-20010028
Record Dates: First submitted 2020-07-01; First posted 2020-07-07 (Actual); Last update posted 2025-04-16 (Actual); Status verified 2025-04

CONDITIONS: Healthy Children
MeSH Terms: interventions — Fish Oils

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (4):
- Milk Drink Unfortified (Negative Control) (Placebo Comparator): Children will get the product (packed for its individual portion) that must be consumed once a day for 30 days.
  Interventions: Dietary Supplement: DHA Wet Mixing method; Dietary Supplement: DHA Dry Blending Method; Dietary Supplement: Fish Oil
- Milk Drink Unfortified Plus Fish Oil (Positive Control) (Active Comparator): Children will get the product (packed for its individual portion) that must be consumed once a day for 30 days
  Interventions: Dietary Supplement: DHA Wet Mixing method; Dietary Supplement: DHA Dry Blending Method
- Milk Drink Fortified with DHA Used Wet Mixing Method (Experimental): Children will get the product (packed for its individual portion) that must be consumed once a day for 30 days
  Interventions: Dietary Supplement: DHA Dry Blending Method; Dietary Supplement: Fish Oil
- Milk Drink Fortified with DHA Used Dry Blending Method (Experimental): Children will get the product (packed for its individual portion) that must be consumed once a day for 30 days
  Interventions: Dietary Supplement: DHA Wet Mixing method; Dietary Supplement: Fish Oil

INTERVENTIONS:
Dietary Supplement: DHA Wet Mixing method — Children will drink milk contain 100 mg DHA wet mixing daily for 30 days
  Arms: Milk Drink Fortified with DHA Used Dry Blending Method; Milk Drink Unfortified (Negative Control); Milk Drink Unfortified Plus Fish Oil (Positive Control)
Dietary Supplement: DHA Dry Blending Method — Children will drink milk contain 100 mg DHA dry blending daily for 30 days
  Arms: Milk Drink Fortified with DHA Used Wet Mixing Method; Milk Drink Unfortified (Negative Control); Milk Drink Unfortified Plus Fish Oil (Positive Control)
Dietary Supplement: Fish Oil — Children will have this intervention every day for 30 days
  Other Names: Children will have milk drink and Fish Oil contain 100 mg/DHA daily for 30 days
  Arms: Milk Drink Fortified with DHA Used Dry Blending Method; Milk Drink Fortified with DHA Used Wet Mixing Method; Milk Drink Unfortified (Negative Control)

SUMMARY:
Infants and young children have high nutritional demands in order to support adequate growth and development, particularly during the transition from complementary feeding at 12 months of age to a mixed and varied diet at 36 months of age. Omega-3 long chain polyunsaturated fatty acid (n-3 LC-PUFA) such as docosahexaenoic acid (DHA; 22:6n-3) is the important constituents of the maturing brain, especially for visual and cognitive development. However only certain foods, such as fatty fish, contain n-3 LC-PUFA at concentrations sufficient for their needs. Additionally, these foods that are known to be rich in DHA may not be regularly provided to infants and toddlers due to concerns about potential food allergies or methylmercury exposure.

Although the importance of consuming n-3 LC-PUFA and essential fatty acids at the level of dietary recommendations in late infancy and early childhood (6-24 months) are highlighted, the current median n-3 LC-PUFA and estimated DHA intakes in toddlers in most countries are lower than the recommended levels. The European Food Safety Authority (EFSA) recommend that infants and young children (< 24 months) should consume 100 mg of DHA per day, while for older children (2-18 years), they recommend a daily intake of 250 mg. In order to bridge the gap between the current intake and recommended levels of n-3 LC-PUFA, general foods, especially infant and toddler formulas, should be enriched with n-3 LC-PUFA particularly DHA. With a growing body of research, the challenge is to find an ideal formula that is nutritionally balanced and human milk-like, especially with respect to the ratio between omega-6 and omega-3 fatty acids and DHA level.

In adding DHA into the toddler formula, there are several methods, among others are in the form of wet mix and dry blending. The aim of this study is to compare the bioavailability of different methods of adding DHA (dry blend versus wet mix) into formulas in healthy Indonesian toddlers age 2-3 years old for a period of one month. Furthermore, to evaluate the stability of milk-based formulas that are supplemented with DHA under same storage conditions, so as to monitor the stability of infant formula.

DETAILED DESCRIPTION:
This study will use two phase approaches Phase 1, screening habitual n3 intake. Mothers of healthy toddlers, non-fish or non-n3 supplement babies (aged 2-3 years old) would be invited to complete a Food Frequency Questionnaire (FFQ) to determine their habitual dietary intake of long chain n3 fatty acids. The 120 babies with the lowest long chain n3 intake would be invited to proceed to phase 2 of the trial.

Phase 2, double blinded, randomized trial. Based on the outcome of the FFQ in phase 1 of the proposed trial, the 120 babies with the lowest habitual dietary intake will be allocated to diet in a random order for one month. Blood samples will be collected via dry blood spot kits at the start, middle and end of the diet along with faecal collection every day.

Groups are Milk drink unfortified (negative control), Milk drink unfortified plus fish oil (positive control), Milk drink fortified with DHA used wet mixing method and Milk drink fortified with DHA used dry blending method.

Population and subjects are Indonesian children aged 2-3 years old living in Jakarta will be selected if they meet the study criteria.

For stage-1: to get 50% of children having habitual low DHA intake, with degree of significance 5% and degree of reliability 95%, then 385 children will be needed.

For stage-2: This study will include 30 subjects per-study group

ELIGIBILITY:
Inclusion Criteria:

* Boys and girls aged 2-3 years old, apparently healthy, living in the study area for minimally one month and parents permit them to participate in the study by signing the informed consent.

Exclusion Criteria:

* Having milk allergy and/or lactose intolerance, high omega-3 intake habit

Ages: 2 Years to 3 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 91 (Actual)
Dates: Start 2023-02-17 (Actual); Primary Completion 2024-03-01 (Actual); Study Completion 2024-05-30 (Actual)

PRIMARY OUTCOMES:
DHA level in RBC lipid and faecal | One month
  Blood and faecal specimen

CONTACTS AND LOCATIONS:
Overall Officials: Diana Sunardi, Doctor, Principal Investigator — Faculty of Medicine University of Indonesia Cipto Mangunkusumo Hospital
Locations (1):
- Sekretariat RW 12 Cipinang besar, Jakarta, DKI Jakarta, Indonesia

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Keim SA, Branum AM. Dietary intake of polyunsaturated fatty acids and fish among US children 12-60 months of age. Matern Child Nutr. 2015 Oct;11(4):987-98. doi: 10.1111/mcn.12077. Epub 2013 Sep 13. PMID 24034437
- [Background] Osendarp, S.J., The role of omega-3 fatty acids in child development. Oléagineux, Corps gras, Lipides, 2011. 18(6): p. 307-313
- [Background] EFSA Panel on Dietetic Products, N.a.A. and Allergies, Scientific Opinion on the substantiation of a health claim related to DHA and contribution to normal brain development pursuant to Article 14 of Regulation (EC) No 1924/2006. EFSA Journal, 2014. 12(10): p. 3840
- [Background] Meyer BJ, Mann NJ, Lewis JL, Milligan GC, Sinclair AJ, Howe PR. Dietary intakes and food sources of omega-6 and omega-3 polyunsaturated fatty acids. Lipids. 2003 Apr;38(4):391-8. doi: 10.1007/s11745-003-1074-0. PMID 12848284
- [Background] Innis SM, Vaghri Z, King DJ. n-6 Docosapentaenoic acid is not a predictor of low docosahexaenoic acid status in Canadian preschool children. Am J Clin Nutr. 2004 Sep;80(3):768-73. doi: 10.1093/ajcn/80.3.768. PMID 15321820
- [Background] Barbarich BN, Willows ND, Wang L, Clandinin MT. Polyunsaturated fatty acids and anthropometric indices of children in rural China. Eur J Clin Nutr. 2006 Sep;60(9):1100-7. doi: 10.1038/sj.ejcn.1602424. Epub 2006 Mar 15. PMID 16538238
- [Background] Kim Y, Kim H, Kwon O. Dietary intake of n-3 and n-6 polyunsaturated fatty acids in Korean toddlers 12-24 months of age with comparison to the dietary recommendations. Nutr Res Pract. 2019 Aug;13(4):344-351. doi: 10.4162/nrp.2019.13.4.344. Epub 2019 Jul 24. PMID 31388411
- [Background] Tsuboyama-Kasaoka N, Takizawa A, Tsubota-Utsugi M, Nakade M, Imai E, Kondo A, Yoshida K, Okuda N, Nishi N, Takimoto H. Dietary intake of nutrients with adequate intake values in the dietary reference intakes for Japanese. J Nutr Sci Vitaminol (Tokyo). 2013;59(6):584-95. doi: 10.3177/jnsv.59.584. PMID 24477258
- [Background] Gibson, S. and A. Sidnell, Nutrient adequacy and imbalance among young children aged 1-3 years in the UK. Nutrition bulletin, 2014. 39(2): p. 172-180